CLINICAL TRIAL: NCT03117647
Title: Is Early Intervention Using Mansoura-VV Uterine Compression Sutures an Effective Procedure in the Management of Primary Atonic Postpartum Hemorrhage? : A Prospective Study
Brief Title: Mansoura-VV Uterine Compression Suture for Primary Atonic Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, WaleedAl Refaie, associate professor, Mansoura University
Other Study IDs: R/16.09.55
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mansoura-VV compression suture — two compression suture both are v shaped apex of each suture placed 2 cm below suture line of C.S and 3 cm from the lateral border of the uterus on the right and left side

SUMMARY:
Postpartum hemorrhage is the leading cause of maternal, uterine atony accounts for 75-90% of primary postpartum hemorrhage. The efficacy of the Uterine compression suture in the treatment of atonic postpartum hemorrhage is time-tested and can be said to be almost established .The aim of this study was to assess the role of the Mansoura-VV uterine compression suture as an early intervention in the management of primary atonic postpartum hemorrhage.

DETAILED DESCRIPTION:
This prospective observational study was carried out at the Obstetrics and Gynecology Department Mansoura University Hospital, and private settings in Mansoura, Egypt, during the period from May 2013 to December 2016. Inclusion criteria included women diagnosed with primary atonic PPH, during cesarean section when the uterus failed to contract after the routine doses of uterotonics. Women and their partners were counseled and signed a consent regarding the technique as an alternative to devascularization or hysterectomy. Exclusion criteria included patients with placenta previa complete or incomplete centrails, and/or placenta accreta. Also one case of atonic PPH, when the uterus was incompressible and failed to contract on bimanual compression was excluded from the study, as in our experience these cases failed to respond to any type of UCS.

In this series, immediately after anesthesia, all women received misoprostol 400 mcg (two tablets of MisotacR, Adwia Co, 6th October city, Egypt) sublingual, as well as 20 IU of oxytocin (Syntocinon, Sanofi Aventais, Egypt) in 50 0-mL lactated Ringer's solution as an intravenous infusion, after delivery of the baby and clamping of the umbilical cord. This is routine practice for all women undergoing CS in our department.

After closure of the uterine incision, uterine atony was diagnosed in 108 women when the uterus felt soft and flappy, and failed to respond to intermittent fundal massage, the second dose of the previously mentioned ecbolics was given. Then, bimanual compression of the uterus was attempted for 10 to 15 minutes until the tone of the uterus is regained as well as to assess the potential chances of success of the Mansoura-VV uterine compression suture.

Within 15 minutes of the diagnosis, the uterus was rechecked to identify any bleeding points. the investigators performed Mansoura-VV uterine compression suture. The right V was performed as follow: (i) 100-cm Vicryl no. 1 was thrown to form two nearly equal parts (each 50 cm) on a blunt semicircular 70-mm needle, the curve of the needle was straightened. (ii) The needle transfixed the right uterine wall from anterior to posterior, about 2 cm below the hysterotomy incision and 3 cm from the (this represents the apex of the V suture). (iii) after transfixation, the Vicryl was divided thus two threads from one transfixation each 50-cm threads penetrated the lower uterine segment; medial (M) and lateral (L) threads, each has anterior (aL and aM) and posterior (pL and pM) ends in relation to the uterus (iv) The free anterior and posterior ends of the lateral thread (aL and pL) were tied above the fundus with three double - throw knots about 3 cm from the right cornual border of the uterus forming the lateral limb of the V suture. (v) The free anterior and posterior ends of the medial threads (aM and pM) were tied above the fundus 2-3 cm medial to the lateral limb completing the V suture . The lead surgeon pulled the suture to provide moderate tension, while the assistant surgeon lift the uterus upward while perform a bimanual uterine compression to minimize trauma and to achieve or aid compression during the ligation of each vertical limb. (vi) using a similar technique, the left V suture was laid on the left side, and then the VV suture is completed.

The vagina was inspected to check for control of bleeding with Mansoura-VV sutures, the uterus cannot be stretched. Only one case (1/108) required additional bilateral uterine vessels ligation for control of bleeding, the abdomen was closed routinely. Antibiotics were given and continued postoperatively for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with atonic postpartum hemorrhage at the time of cesarean section after appropriate use of ecobolics

Exclusion Criteria:

* patients with placenta previa complete or incomplete centrails, and/or placenta accreta

Ages: 19 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: women diagnosed with primary atonic PPH, during cesarean section when the uterus failed to contract after the routine doses of uterotonics.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
primary postpartum haemorrhage from atony | first 24 hours post partum
  blood loss more than 1000 cc.

REFERENCES:
- [Derived] El Refaeey AEA, Abdelfattah H, Mosbah A, Gamal AM, Fayla E, Refaie W, Zaied A, Barakat RI, Seleem AK, Maher M. Is early intervention using Mansoura-VV uterine compression sutures an effective procedure in the management of primary atonic postpartum hemorrhage? : a prospective study. BMC Pregnancy Childbirth. 2017 May 31;17(1):160. doi: 10.1186/s12884-017-1349-x. PMID 28569213